CLINICAL TRIAL: NCT06634862
Title: Comparison of the Effects of Intermittent Pneumatic Compression, Graston Technique and Percussive Therapy on Muscle Pain, Muscle Tone and Balance After Quadriceps Fatigue Protocol
Brief Title: Comparison of the Effects of Intermittent Pneumatic Compression, Graston Technique and Percussive Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Melis Beril Yazıcı, Master of Science, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-FTR-MBY-01
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Recovery Method
Keywords: Recovery; Quadriceps Fatigue Protocol; Intermittent pneumatic pressure; Soft Tissue Mobilization Technique; Percussive therapy; Muscle Fatigue; Muscle Tone

STUDY DESIGN:
Intervention Model Description: Four groups, together with a control group with no intervention. One group will receive pneumatic pressure treatment, one group will receive soft tissue mobilisation (graston) treatment and another group will receive percussive therapy treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- intermittent pneumatic pressure group (Other): Intermittent Pneumatic Compression (IPC) is a mechanical method of applying compression to the limbs and has a number of therapeutic uses. The device consists of a pair of inflatable sleeves wrapped around the leg and an electric pneumatic pump that inflates the sleeves with air, compressing the deep veins and displacing blood proximally. The working principle of IPC is based on passively increasing blood flow by applying external pressure to the extremity, but the exact physiological mechanisms are only partially understood. However, despite its widely recognised use and positive effects on circulatory conditions, the literature on the use of IPC in musculoskeletal treatment is limited. The available evidence has been investigated in several studies, including the efficacy of IPC, its effect on vasodilatory effects in distal skeletal muscle and its effect on serum indices of muscle function, pain and muscle damage. Studies have also reported improvements in exercise duration as wel
  Interventions: Other: Normatec Air Compression
- Soft Tissue Mobilization Technique Group (Other): The Graston Technique (GT) is a form of instrument-assisted soft tissue mobilisation that uses stainless steel instruments to perform manual therapy on soft tissues. It is widely used by clinicians to treat various soft tissue disorders. Research has reported that it effectively promotes the inhibition of adhesion of treated tissues and collagen synthesis. Furthermore, the graston technique has been used to manage pain and range of motion limitations caused by scar tissue and musculoskeletal injuries. Overall, the graston technique has been studied in a variety of contexts and has demonstrated potential effects on range of motion, pain relief and musculoskeletal conditions. Some studies reported direct effects on specific outcomes, while others emphasised its potential when combined with other therapeutic interventions. These findings contribute to the understanding of the graston technique as a modality for soft tissue mobilisation and musculoskeletal disorders in the field of physio
  Interventions: Other: Soft Tissue Mobilization
- Percussive Therapy Group (Other): Percussive therapy has gained popularity in recent years as a potential intervention to alleviate muscle soreness and fatigue after exercise. This therapy involves the use of a mechanical system to provide percussive massage and its effectiveness in promoting recovery and reducing muscle soreness has been a topic of interest in the field of sports medicine and rehabilitation. Several studies have investigated the acute effects of percussive therapy on muscle recovery and pain, aiming to understand its potential benefits for athletes and individuals engaged in physical activities. Furthermore, the use of percussive therapy with resistance training has been shown to have acute effects on movement speed, suggesting the potential to influence exercise performance and recovery. These findings contribute to the understanding of how percussive therapy can influence muscle function and recovery processes. In the context of pain management, exercise therapy is advocated as an effective treatm
  Interventions: Other: Percussive therapy
- control group (No Intervention): In the control group, quadriceps fatigue protocol was applied, measurements were taken on two separate days and no intervention was made.

INTERVENTIONS:
Other: Normatec Air Compression — Intermittent pneumatic pressure has been used in other studies, usually for deep vein thrombosis and vascular disorders. In this way, it has not been compared with other recovery interventions for post-exercise recovery applications.
  Arms: intermittent pneumatic pressure group
Other: Soft Tissue Mobilization — The soft tissue mobilisation technique has been investigated in other studies in terms of its effect on soft tissue and its role recovery. In this way, there is no comparison with other recovery interventions for post-exercise recovery applications.
  Arms: Soft Tissue Mobilization Technique Group
Other: Percussive therapy — Percussive therapy has been investigated in device research and athlete health. In this way, it has not been compared with other recovery interventions for post-exercise recovery applications.
  Arms: Percussive Therapy Group

SUMMARY:
The aim of this study was to compare the effects of intermittent pneumatic pressure, percussive therapy and graston after a fatigue protocol applied to the leg muscles.

DETAILED DESCRIPTION:
a- Subject and Objective (the importance of the subject, why this subject is the problem and the objectives of the study will be written based on the literature with the narration of the researcher):

Studies on the intermittent pneumatic compression device, graston technique and percussive therapy (massage weapons) have focused on investigating their use in athlete health. During the literature review, it was realised that the use of these and other auxiliary therapies and elements that increase the speed of recovery has not been investigated for sedentary individuals. The necessity and benefits of regular exercise for sedentary individuals as well as athletes in daily life have been proven by many studies. It has become a common belief that exercise should be a part of the life of every adult individual, whether athlete or sedentary, in order to maintain a healthy life. Furthermore, enjoyment of exercise and perceived exercise intensity play an important role in the adherence of sedentary individuals; moderate intensity exercise is more likely to be enjoyable and adaptive for this population. Psychological factors such as mood and self-efficacy also influence exercise behaviours in sedentary individuals, with negative exercise-related cognitions potentially moderating the exercise-effect relationship and affecting feelings of pleasure during and after exercise. However, one of the biggest obstacles for sedentary individuals to form a sports habit is the fatigue and muscle pain they experience after exercise. These effects, which make it difficult to continue daily life the next day, distract the person from the habit of exercising regularly. Furthermore, the psychosocial benefits of incorporating regular exercise into the daily life flow are well documented and emphasise the wider positive impact of exercise beyond physical health.

Intermittent Pneumatic Compression (IPC) is a mechanical method used to apply compression to limbs and has a number of therapeutic uses. The device consists of a pair of inflatable sleeves wrapped around the leg and an electric pneumatic pump that inflates the sleeves with air, compressing deep veins and displacing blood proximally. The working principle of IPC is based on passively increasing blood flow by applying external pressure to the extremity, but the exact physiological mechanisms are only partially understood. However, despite its widely recognised use and positive effects on circulatory conditions, the literature on the use of IPC in musculoskeletal treatment is limited. The available evidence has been investigated in several studies, including the efficacy of IPC, its effect on vasodilatory effects in distal skeletal muscle and its effect on serum indices of muscle function, pain and muscle damage. Studies have also reported improvements in exercise duration as well as fatigue when using pneumatic compression during rest after warm-up exercises. IPC devices are particularly popular among endurance athletes because they have the potential to reduce exercise-induced muscle damage. Research on IPC has shown that the devices increase muscle blood flow during exercise and increase blood flow during post-exercise recovery. More research is needed on the effects of IPC in musculoskeletal treatment, especially on exercise-induced muscle damage and pain. In conclusion, IPC devices have shown promising results in various therapeutic applications, especially in athlete rehabilitation and post-exercise recovery. Furthermore, all of this information demonstrates the great potential of these devices for health and sports applications.

The Graston Technique (GT) is a form of instrument-assisted soft tissue mobilisation that uses stainless steel instruments to perform manual therapy on soft tissues. It is widely used by clinicians to treat various soft tissue disorders. Research has reported that it effectively promotes collagen synthesis and inhibition of adhesion of treated tissues. Furthermore, the graston technique has been used to manage pain and range of motion limitations caused by scar tissue and musculoskeletal injuries. Overall, the graston technique has been studied in a variety of contexts and has demonstrated potential effects on range of motion, pain relief and musculoskeletal conditions. Some studies reported direct effects on specific outcomes, while others emphasised its potential when combined with other therapeutic interventions. These findings contribute to the understanding of the graston technique as a modality for soft tissue mobilisation and musculoskeletal disorders in the field of physiotherapy and rehabilitation, particularly highlighting its potential to manage muscle pain and promote recovery. In conclusion, the graston technique is a widely used form of instrument-assisted soft tissue mobilisation with reported efficacy in the management of various musculoskeletal disorders.

Percussive therapy has gained popularity in recent years as a potential intervention to alleviate post-exercise muscle pain and fatigue. This therapy involves the use of a mechanical system to provide percussive massage and its effectiveness in promoting recovery and reducing muscle soreness has been a topic of interest in the field of sports medicine and rehabilitation. Several studies have investigated the acute effects of percussive therapy on muscle recovery and pain, aiming to understand its potential benefits for athletes and individuals engaged in physical activities. Furthermore, the use of percussive therapy with resistance training has been shown to have acute effects on movement velocity, suggesting the potential to influence exercise performance and recovery. These findings contribute to the understanding of how percussive therapy can influence muscle function and recovery processes. In the context of pain management, exercise therapy has been advocated as an effective treatment for chronic low back pain, suggesting the potential for therapeutic interventions, including percussive therapy, to address musculoskeletal pain and discomfort. Although the acute effects of percussive therapy on muscle recovery have been the focus of research, the underlying mechanisms and long-term effects of this therapy need to be further investigated. Understanding the impact of percussive therapy on muscle regeneration, inflammation and tissue repair processes may provide valuable insights into its potential to enhance recovery and reduce muscle fatigue. In conclusion, research on massage gun or percussive therapy demonstrates its potential as a valuable intervention to address post-exercise muscle pain and fatigue. Further investigation of the underlying mechanisms, long-term effects and comparative effectiveness of percussive therapy may provide valuable insights into its role in promoting muscle recovery and enhancing exercise performance.

Considering all these, it is necessary to compare these modalities among each other and to investigate their contribution to the health of sedentary individuals as well as athletes. Although there are studies in the literature on the comparison of these modalities with classical physiotherapy and rehabilitation modalities, there is no comparative study on their contribution to the recovery process. In addition to its contribution to the literature, this study is thought to be useful for physiotherapists who use these and similar modalities in the clinical environment.

The main aim of this study was to investigate the effects of these therapeutic treatment modalities on post-exercise muscle pain, muscle tone and fatigue. Post-exercise recovery is a very popular topic in recent times, especially for athletes. Many different methods are used for this purpose in the clinical environment. In this study, the effectiveness of these modalities on recovery and their superiority over each other will be investigated.

H0 Hypothesis: Intermittent pneumatic compression, graston technique and percussive therapy have no effect on muscle pain, muscle tone and balance after quadriceps fatigue protocol.

H1 Hypothesis: Intermittent pneumatic compression device application is more effective than graston technique and percussive therapy on muscle pain, muscle tone and balance after quadriceps fatigue protocol.

H2 Hypothesis: Graston technique application is more effective than intermittent pneumatic compression device and percussive therapy on muscle pain, muscle tone and balance after quadriceps fatigue protocol.

H3 Hypothesis: Percussive therapy is more effective than intermittent pneumatic compression device and graston technique on muscle pain, muscle tone and balance after quadriceps fatigue protocol.

ELIGIBILITY:
Inclusion Criteria:

* To be between 25-45 years old.
* Not having any chronic disease.
* Not doing active sports for at least 6 months.
* Not having any previously diagnosed lower extremity pathology.
* Not having a chronic lower extremity problem and not having a major trauma (fracture, anterior cruciate ligament injury, etc.).
* Not having any cognitive problem that prevents them from following and adapting to a specific exercise programme.
* No visual, vestibular and neurological disorders.

Exclusion Criteria:

* Having a chronic disease.
* Any musculoskeletal problem in the lower extremities.
* Use of sedative medication due to chronic disease (rheumatism, lung and/or heart etc.)
* Regular use of painkillers, muscle relaxants or anti-inflammatory drugs.
* Any history of surgery on the lower extremity.
* Any history of pain in the lower extremity during the fatigue protocol.
* Pregnancy.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-03-16 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Star Balance Test | The balance test will take 10 minutes in total before and after the intervention.
  On the floor, 4 strips of adhesive tape, previously cut 2 metres long, will be glued in such a way that they form 45 degree angles between them. The participant will align in the centre of the star and perform the reaching on one leg in anterior, anteromedial, anterolateral, posterior posterolateral, posteromedial, medial and lateral directions. The test will be performed anti-clockwise if the participant's initial leg is right and the participant will reach with the left leg; clockwise if the initial leg is left and the participant will reach with the right leg. During the test, the participant will be asked to keep his/her hands on his/her waist and not to change his/her position throughout the test. Then the participant will be asked to reach to the last point he/she can reach, touch his/her toe to the strip and return to the starting position. Then he/she will be asked to move to the other line in the specified direction and complete a total of 8 lines in this way.
Muscle pain measurement with algometer | It will take 30 minutes in total before and after the intervention.
  Pressure-pain threshold (PPT) will be measured with a hand-held pressure algometer. The participant will be comfortably seated in an ordinary chair with an adjustable seat and backrest and arms resting on a soft support placed on either side of the chair. The chair height and arm rests will be adjusted so that the subject's knees and hips are in 90° flexion. Two sites/muscles will be marked for use in PPT determinations to avoid peripheral sensitisation due to frequent, multiple PPT assessments at the same site. In M. quadriceps femoris, a site 2.5 cm proximal and 2.5 cm distal to the midpoint between the apex patella and groin will be marked bilaterally. The researcher will instruct the participants to press the button on their own as soon as the pressure sensation becomes painful. The rate of pressure increase of the device will be kept between approximately 40-60kPa.
Muscle tone measurement with MyotonPRO | It will take 30 minutes in total before and after the intervention.
  Measurements of bilateral rectus femoris muscles will be taken twice on the same day and time of the week, one week apart.The first measurement will be made without any intervention and the second measurement will be made after the protocol has been implemented.The test lead of the MyotonPRO will be placed on the skin over the area perpendicular to the surface of the muscle belly and the device will then be placed in the measurement position and held steady while the device automatically performs a series of predefined measurements.The device will be used in multiscan mode, where a measurement consists of the average of 10 mechanical touches one second apart. In the control group and in the first measurement of the experimental groups, the measurement will be performed after the participant has rested for 15 minutes after the fatigue protocol as described above.The second measurement in the experimental groups will be performed as described above without resting after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When the study is finalised, researchers who want to use my data can send me an e-mail and use my data.

REFERENCES:
- [Background] Stedge HL, Armstrong K. The Effects of Intermittent Pneumatic Compression on the Reduction of Exercise-Induced Muscle Damage in Endurance Athletes: A Critically Appraised Topic. J Sport Rehabil. 2021 Jan 8;30(4):668-671. doi: 10.1123/jsr.2020-0364. PMID 33418535
- [Background] Machado AF, Ferreira PH, Micheletti JK, de Almeida AC, Lemes IR, Vanderlei FM, Netto Junior J, Pastre CM. Can Water Temperature and Immersion Time Influence the Effect of Cold Water Immersion on Muscle Soreness? A Systematic Review and Meta-Analysis. Sports Med. 2016 Apr;46(4):503-14. doi: 10.1007/s40279-015-0431-7. PMID 26581833